CLINICAL TRIAL: NCT02396186
Title: An Assessment of the Glider Balloon in Complex Lesions
Acronym: ANTELOPE
Status: Completed | Type: Observational
Sponsor: TriReme Medical, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP785
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PTCA Balloon Angioplasty

SUMMARY:
The purpose of this study is to collect data from real-world use with the Glider Percutaneous Transluminal Coronary Angioplasty (PTCA) Balloon Catheter to support the effectiveness of the Glider PTCA Balloon for crossing into complex coronary lesions.

DETAILED DESCRIPTION:
Observational Study collecting data on commercial cases in which the Glider PTCA Balloon Catheter is used in accordance with the instructions for use. This study includes up 500 patients at up to 50 study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Lesion must be successfully crossed with a guidewire without complication (including Chronic Total Occlusions (CTOs))
2. The Glider balloon may only be used at one lesion during the procedure
3. The lesion in which the Glider balloon is used must be completed first
4. The primary lesion treated during the procedure must be treated with the Glider balloon
5. Intended treatment of a protocol-defined complex lesion that has at least one of the following factors:

   * Significant vessel tortuosity
   * Failed balloon crossing with another balloon
   * Tight stenosis
   * Heavy calcification
   * Side branch present

Exclusion Criteria:

1. Patient < 18 years of age
2. Lesion longer than 40mm
3. Device use not consistent with Instructions for Use
4. Patient has not given consent for their data to be submitted to this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of coronary interventions involving the Glider™ PTCA Balloon Catheter at participating centers will be reviewed for patient eligibility. Patients from all eligible cases should be invited to sign an IRB-approved Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Technical Success Rate | 1 hour
  Percentage of lesions successfully crossed among those attempted with the Glider PTCA catheter.

SECONDARY OUTCOMES:
Freedom from Balloon Slippage | 1 hour
  Percentage of inflations with the Glider balloon in which the physician user reports no slippage.
Lesion Success Rate | 48 hours
  Percentage of lesions with <50% diameter stenosis, or Thrombolysis In Myocardial Infarction (TIMI) 3 flow if side branch is present, without development of MACE during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: David Rizik, MD, Principal Investigator — Scottsdale Healthcare; William Lombardi, MD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Alexian Brothers Heart and Vascualr Institute, Elk Grove Village, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - York Hospital, York, Pennsylvania
  - Cardiovascular Specialists of Texas, Austin, Texas